CLINICAL TRIAL: NCT04469257
Title: THE EFFECT OF SUN LIGHT EXPOSURE TO THE LEVEL OF VITAMIN D IN THE ELDERLY LIVING IN NURSING HOME
Brief Title: SUN LIGHT EXPOSURE AND VITAMIN D LEVEL IN NURSING HOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Fatih OKAN, LECTURER PHD., Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 123457
Record Dates: First submitted 2020-07-06; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Nursing Home; Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Intervention Model Description: pretest-posttest randomized controlled experimental study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sunbathing (Experimental): During the activities for the intervention group, the individuals were exposed directly to sun in the nursing home garden on open and sunny days without sunscreen for five days a week for a month with an average of 21.0 ± 5.0 min (min 15 min - max 30 min). About 30-35% of their bodies (hand, face, neck, forearm open up to elbows and legs open up to the knee caps) were open. Sunbathing sessions were held between 10:30 and 11:30 to prevent elderly individuals from being affected by extreme temperatures, and UV index values were monitored during the time and duration of the event at WHO website (http://www.who.int/uv/resources/link/indexlinks/en/, Access date: July 1, 2018). During the hours of the day when UV index was > 6-7, elderly individuals were not taken out. After each sunbathing session, elderly individuals in the intervention group were evaluated for sensitivity and erythema that may occur in the exposed body areas
  Interventions: Behavioral: Sunbathing
- Control (No Intervention): Elderly individuals in the control group were not invited to the activities held in the nursing home garden. There were no restrictions on them for not going out in the sun or spending time inside the nursing home

INTERVENTIONS:
Behavioral: Sunbathing — the individuals were exposed directly to sun in the nursing home garden on open and sunny days without sunscreen for five days a week for a month with an average of 21.0 ± 5.0 min (min 15 min - max 30 min). About 30-35% of their bodies (hand, face, neck, forearm open up to elbows and legs open up to the knee caps) were open.
  Arms: Sunbathing

SUMMARY:
Objective: The aim of the present study was to determine the effect of nursing interventions and sunlight exposure to reach optimum vitamin D levels by individuals living in nursing homes on vitamin D levels.

Material Method: In the first stage of this two-stage randomized-controlled experimental study with pretest-posttest design conducted in June - August 2018 period in the nursing home in Central Town of Tokat Province, the questionnaire prepared by the researcher, standardized mini mental test, Fitzpatrick skin typing questionnaire and Katz Index of activities of daily living were applied. Intervention (n=20) and control (n=20) groups were established with individuals using simple random method according to age, gender, skin type and vitamin D level. In the second stage, 30-35% of the body surface area of individuals in the intervention group was exposed to sunlight five days a week in July. For the participants in the control group, sunbathing was not offered. 25(OH)D, calcium, parathormone, phosphorus, alkaline phosphatase and albumin levels of all individuals were measured in blood samples taken at the beginning and end of the study. Two-way mixed ANOVA, Mann-Whitney U test, Wilcoxon signed rank test and Chi-square tests were used to evaluate the data.

ELIGIBILITY:
Inclusion Criteria:

* individuals (25 women and 41 men) who lived in nursing home during June 27, 2018 and August 01, 2018 period
* 60 years and older
* able to perform their daily life activities independently
* agreed to participate in the study

Exclusion Criteria:

* malignancies
* advanced liver and kidney failure
* history of gastric-bowel operation
* skin disease that could prevent sun exposure
* hyperparathyroidism
* malabsorption
* use of drugs that affect the levels of vitamin D, calcium, PTH and phosphorus and albumin

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Vitamin D | 5 week
  Vitamin D Level

SECONDARY OUTCOMES:
Parathormone | 5 week
  Parathormone level
Calicium | 5 week
  Calcium Level
Phosphorus | 5 week
  Phosphorus level
Alkaline Phosphatase | 5 week
  Alkaline phosphatase level
Albumin | 5 week
  Albumin level

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No